CLINICAL TRIAL: NCT00289380
Title: 1. Prevalence of Nutritional Risk-undernutrition-support in China-Euro-USA. 2. Impact of Nutrition Support on Outcome for Patient at Risk. 3. Impact of Nutrition Support on Outcome,Cost/Effectiveness for Patient at Risk.
Brief Title: Nutrition Support on Outcomes and Cost-effectiveness for Patients at Risk
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Zhu-ming Jiang, Professor of General Surgery,, Peking Union Medical College
Other Study IDs: CMA2005CSPEN
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Malnutrition; Nutritional Risk
Keywords: Nutritional Risk Screening(NRS); Malnutrition; Overweight; Obesity; Clinical nutritional support; Clinical outcome; Cost effectiveness; Complication; Infective complications
MeSH Terms: conditions — Malnutrition; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Nutrition support: Nutrition support cohort means accept nutrition support，it was defined as ≥15kal/kg/d and < 30kal/kg/d of non-protein calories (carbohydrate and/or fat) and amino acids or protein≥1g/kg/d for 5~28 consecutive days.
- Without nutritional support: Group received only intravenous 5 to 10% glucose and electrolyte infusions

SUMMARY:
1. The aim of this large scale study to survey the prevalence of nutritional risk and malnutrition in China,Europe and USA.
2. The impact of nutritional support for the patients at nutritional risk on clinical outcomes and cost-effectiveness

Already get the approval by Ethics Committee of Peking Union medical college and Johns Hopkins Hospital.

DETAILED DESCRIPTION:
Although it was often to hear that malnutrition ratio in Aisa hospitalized patient was 40%-70% , there was no evidence to elaborate the prevalence of nutritional risk and malnutrition on hospitalized patients of Asia. Also in USA no data for nutritional risk. In 2002, scientists group headed by Kondrup from : European Society for Parenteral and Enteral Nutrition demonstrated that randomized controlled clinical trials showed patients may get benefit from nutrition support when they with nutrition risk. Based on these evidences, a simpler method was established by European Society for Parenteral and Enteral Nutrition in year 2002 in Munich & it was demonstrated useful to evaluate the appropriate use of nutrition support at present time. This method was named as Nutrition Risk Screening (NRS).

We propose to survey the prevalence of malnutrition & nutrition risk in large cities' large/middle size hospitalized patients in China, Europe and USA use NRS tool. As well, we also aim to figure out the current nutrition support status in current large/middle size hospitals through this survey.

we also propose to evaluate the cost-effectiveness of parenteral nutrition, enteral nutrition and non-nutritional support, and to examine the clinical outcomes of nutritional support in certain patients at nutritional risk identified by NRS-2002.

For international cooperation,our partners are Professor Kondrup of Europe and Professor Nolan from Johns Hopkins Hospital,there are students from a cooperative project with Johns Hopkins Hospital for Doctor of Philosophy students 2005-2011.

In plan this protocol might be completed around 2016 also.

ELIGIBILITY:
Inclusion Criteria:

* patients be in hospital overnight
* diagnoses according to the protocol of cohort study for cost effectiveness

Exclusion Criteria:

* patients admitting from emergency department
* patients who undergone operation before second morning of hospitalization
* patients who dose not give Informed Consents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuing sampling in 6 clinical Departments of large, middle & small size hospitals in 15 large cities from West, Middle & East China.
  Also, data from Denmark and USA will be collected and analysed.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2005-01; Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Infectious complication | Observation will be carried from admitting end until discharge
  A infectious complication was defined as as the presence of recognized pathogens in body tissues that normally are sterile, confirmed by the results of culture and supported by clinical, radiologic or hematologic evidence of infection

SECONDARY OUTCOMES:
cost effectiveness | Observation will be carried from admitting end until discharge
  The cost effectiveness analysis was performed from the payers' perspective.The percentage of infectious complication-free patients was used to measure the effectiveness. The total cost was considered to contain 3 items in our study. The first item was the cost of nutrition support, including nutrition solutions, nursing, physician, and other staff supervision of nutrition support preparation, administration, and catheter placement and maintenance. The second item was the cost of the infectious complication.The third item was 'other costs' associated with the hospital admission, calculated from the total costs from which the cost of nutrition support and infectious complications were subtracted. The incremental cost-effectiveness ratio (ICER) was calculated by dividing the costs difference between the nutrition support cohort and no-nutrition support cohort by their difference in effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu-ming Jiang, M.D., FACS, Study Director — Peking Union Medical College Hospital
Locations (15):
- China (15):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Medical Univ. Hospital, Chongqing, Chongqing Municipality
  - Xin Qiao Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospial, Guangxi Medical University, Nanning, Guangxi
  - The First University Hospital, Hebei Medical University, Shijiazhuang, Hebei
  - Nankai Hospital, Tianjin, Hebei
  - Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - Xin Hua Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Sixth Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Xinjiang Medical University, Ürümqi, Xinjiang
  - Second Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Jie B, Jiang ZM, Nolan MT, Efron DT, Zhu SN, Yu K, Kondrup J. Impact of nutritional support on clinical outcome in patients at nutritional risk: a multicenter, prospective cohort study in Baltimore and Beijing teaching hospitals. Nutrition. 2010 Nov-Dec;26(11-12):1088-93. doi: 10.1016/j.nut.2009.08.027. Epub 2009 Dec 5. PMID 19963351